CLINICAL TRIAL: NCT03491254
Title: A Multisite, Open-label, Prospective Cohort Study Investigating Huaier Granule Combined With Biliary Drainage for Treatment of Malignant Obstructive Jaundice（MOJ）
Brief Title: Investigating the Efficacy and Safety of the Combination Treatment of Huaier Granule and Biliary Drainage for MOJ
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: zhaoyu liu (Other)
Responsible Party: Sponsor-Investigator, zhaoyu liu, Professor, Shengjing Hospital
Organization: Shengjing Hospital (Other)
Other Study IDs: HE-201801
Record Dates: First submitted 2018-03-22; First posted 2018-04-09 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Obstructive Jaundice
MeSH Terms: conditions — Jaundice, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A/exposure group: Huaier Granule & biliary drainage
- Group B/non-exposure group: biliary drainage.

SUMMARY:
This study is designed to evaluate the efficacy and safety of the combination treatment of Huaier granule and biliary drainage for malignant obstructive jaundice.

DETAILED DESCRIPTION:
After sign the informed consent, the, eligible patients are those who have completed the examinations within 2 weeks after the biliary drainage will enter the study and visit the study sites at Weeks 12, 24, 36, and 48. The follow-up duration is up to 48 weeks or until the death of patient during the study. The patients will be allocated to two groups based on whether being exposed to Huaier granule or not.

Study data will be collected prospectively, including the patients' baseline characteristics, chemo-/radio-therapy history, previous Huaier granule treatment, laboratory tests, imaging examinations, and various clinical endpoints including liver function, quality of life, status of survival, and safety.

This is a non-interventional study in patient population in real world. Therefore, the patients' treatment regimen will not be interfered, i.e., the patients will independently decide whether to take Huaier granule or not based on the recommendation from the clinician after the drainage. The patients will be allocated into different groups completely according to their treatment at clinic in real world. During the study, only the study required data and endpoints will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged between 18~75 years;
2. Naïve patients who were diagnosed as malignant obstructive jaundice that was caused by carcinoma of head of pancreas, cholangiocarcinoma, gallbladder carcinoma, or duodenal papilla carcinoma, or carcinoma metastasis in hilar lymph nodes based on clinical assessments and/or pathological examination;
3. Total bilirubin >80 umol/L;
4. Patients who are not indicated for or refused to receive surgical resection;
5. ECOG score ≤2 or KPS score ≥60;
6. Expected survival time ≥12 weeks;
7. Has signed and dated the informed consent in volunteer and are willing to comply with the data collection procedures by Investigator.

Exclusion Criteria:

1. Female patients who are pregnant or breastfeeding;
2. Patients who are receiving concomitant intravenous chemotherapy;
3. Patients whose malignant obstructive jaundice was caused by liver cancer;
4. Patients who have severe coagulation disorders and massive ascites;
5. Patients with obstructive jaundice who have concomitant fever;
6. Patients who are not applicable for or not willing to receive biliary drainage;
7. Patients who are not appropriate to participate in the study at discretion of the Investigator.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with malignant obstructive jaundice
Sampling Method: Non-Probability Sample
Enrollment: 852 (Estimated)
Dates: Start 2018-05-30 (Estimated); Primary Completion 2020-11-30 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | every 12 weeks until death, up to 48 weeks
  the time interval between baseline and the time of death due to any cause

SECONDARY OUTCOMES:
overall survival rate | 48 weeks
  Overall survival rate at 48 weeks was defined as the proportion of patients who were alive at 48 weeks
Median survival time (MST) | 48 weeks
  indicate the survival time when only 50% of patients are still alive.
Karnofsky (KPS) score | 48 weeks
  improved is defined as KPS increases >10 after treatment; worsen is defined as KPS decreases >10; stable is defined as KPS changes ≤10.
Liver function 1 | 12、24、36、48 weeks
  Measurement of direct bilirubin
Liver function 2 | 12、24、36、48 weeks
  Measurement of total bilirubin
Liver function 3 | 12、24、36、48 weeks
  the time of reoccurrence of jaundice.
Quality of Life (QoL) score | 48 weeks
  Quality of Life (QOL) were measured using supplemental quality of life questions. Item score range（12 items）: 1(worst symptom) to 5 (no symptom). Change: score at 48 weeks minus score at baseline.
Adverse Events | 12、24、36、48 weeks
  Incidence rate of Adverse events